CLINICAL TRIAL: NCT02898883
Title: Building Resilience After Childhood Emergencies (BRACE): A Randomized Trial Examining Efficacy and Feasibility
Brief Title: Building Resilience After Childhood Emergencies (BRACE)
Acronym: BRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Akron Children's Hospital (Other); Kent State University (Other)
Responsible Party: Principal Investigator, Norah Feeny, Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BRACE
Record Dates: First submitted 2016-08-24; First posted 2016-09-13 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Early intervention Program The early intervention program (EIP) will consist of 4 sessions with one parent/guardian of the injured child and a clinical psychology graduate student therapist. All sessions are one on one for one hour. The first session will be conducted in the hospital within an average of 24- 48 hours after the traumatic event. The subsequent three sessions will be conducted electronically via web-based video chat once per week. In general, the EIP will utilize psychoeducation, skills implementation, and daily monitoring to facilitate communication regarding the traumatic event, maintain daily and sleep routines, increase child's access to social support and mitigate the impact of life stress.
  Interventions: Behavioral: Building Resilience after Childhood Emergencies (BRACE)
- Treatment as Usual (TAU) (No Intervention): As part of routine hospital protocol, all participants who screen positively for PTSD risk are provided with a packet of educational materials and potential referrals for behavioral healthcare.

INTERVENTIONS:
Behavioral: Building Resilience after Childhood Emergencies (BRACE) — See arm/group description for details regarding this intervention
  Arms: Intervention group

SUMMARY:
The investigators study seeks to evaluate the feasibility and efficacy of a parent-focused, early intervention to prevent the development of chronic PTSD for children admitted to the emergency department for an acute traumatic injury and their parents. Furthermore, the investigators will identify potential risk factors for the development of PTSD and factors that influence treatment response. Finally, the investigators will prospectively measure trajectories of parental and child responses to trauma and their interaction over time. This study will bring together a multidisciplinary team across two major research universities (Case Western Reserve University and Kent State University) and a large pediatric trauma center (Akron Children's Hospital) in an effort to reduce rates of PTSD in children following traumatic injury.

DETAILED DESCRIPTION:
Objectives:

The proposed research study will evaluate the feasibility and efficacy of an early parent-focused intervention to prevent the development of PTSD for children admitted to the hospital after suffering a medical injury who are at-risk of developing PTSD. Children presenting to the ED with injuries sufficient to warrant admission to the hospital (see below for criteria for trauma admissions), who show risk for PTSD according to a standardized assessment and their parents will be approached to participate in the study. After consenting/assenting to participate in research, children and parents will be randomized to receive the study intervention or treatment as usual. The primary goal will be to measure differences between the study groups on PTSD diagnosis and severity at 1-. 3-, and 6-months post trauma, as well as differences in comorbid diagnoses (e.g., depression), global/scholastic functioning, and other domains targeted by the intervention (e.g., sleep quality, life stress, and social support). The secondary goal will be to measure the impact of parental/ family factors (e.g., parental pathology and family stressors) on children's trajectories of pathology and resilience. The final goal will be to identify salient changes in methylation levels for both parent and child after trauma and the relationship of those changes with the development of symptoms or maladaptive coping. The study will bring together a multidisciplinary team of medical and psychological professionals to build upon a growing literature supporting the use of targeted early interventions to prevent PTSD.

Specific Aims and Hypotheses:

1. Determine the preliminary efficacy of a parent-focused, early intervention to prevent the development of chronic PTSD and other trauma-related outcomes in children exposed to acute, traumatic injury, and their parents. Outcomes will be measured by child self-report, parental self-report, and parental report of the child at intake and follow-up assessments (1-, 3-, and 6-months post trauma). It is hypothesized that the treatment group (early intervention) will show significantly lower rates of PTSD symptoms and associated markers of psychological functioning and higher well-being at all follow-up assessments compared to the treatment as usual (TAU) group. Also, child and parent factors will predict the development of PTSD and treatment response. Finally, the slope of symptom change for parents and their children will be related across time in both groups, and that the slope of symptom change will be moderated by treatment group, with parents and children who received treatment showing greater reductions in symptoms over time.
2. Evaluate the feasibility of a parent-focused, early intervention to prevent the development of chronic PTSD in children exposed to acute, traumatic injury. Feasibility will be determined by participant enrollment and dropout rates, as well as participant subjective ratings of satisfaction with their treatment. It is hypothesized that the intervention will be well-received by participants and that participant enrollment goals will be met.
3. Understand the trajectory of epigenetics (through methylation levels) after a trauma and the relationship between methylation levels and psychological functioning for both parents and children. The investigators will also, investigate the impact of an early intervention on epigenetics in parents and children exposed to an acute injury.

Study Design:

The proposed study will utilize a longitudinal design to measure the effect of early intervention to prevent the development of PTSD symptoms in children (and their parents) exposed to acute traumatic injury. Parent/child dyads entering the study will have an initial assessment after admission to the hospital, within approximately 24-48 hours after the trauma. CHMCA follows recommendations of the American College of Surgeons Committee on Trauma in determining whether a patient's injuries are sufficient to necessitate a trauma admission. Criteria for activating a Trauma Team response are either physiologic (based on HR, blood pressure, mental status, etc) or anatomic (based on extent of identified injuries, such as presence of fractures, penetrating injuries of the torso/head, chest wall injuries, etc), or a combination of the two. Once a trauma team is called, patients are typically admitted for a minimum of 15 hours. As part of the trauma admission process, patients will be screened for PTSD severity using the STEPP. PTSD risk based on this measure is one of the inclusion criteria for this study.Those enrolled in the study will be assigned to 4 sessions of an early intervention or a treatment as usual group. Parent/child dyads will then be assessed again at 1 month, 3 months and 6 months post-trauma. The longitudinal design will allow for the prospective measurement of the effect of predictive factors on the development of PTSD and treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be between the ages of 8 and 13
* Patient must be admitted to the hospital as a trauma admission due to their traumatic injury
* Patient must be accompanied by a legal guardian
* Patient must meet threshold for risk of PTSD
* Both patient and parent must be fluent in English

Exclusion Criteria:

* Intellectual disability or brain damage
* Lower than a 14 on the Glasgow Coma Scale
* Patients who are not deemed sufficiently medically stable to participate by their designated attending physician
* Patients or parents who arrive at the ED intoxicated
* Patients who are not alert, oriented, coherent, or capable of responding to questions

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
UCLA Posttraumatic Stress Disorder Reaction Index (UCLA-PTSD-RI) | 1 month post baseline
  Child PTSD severity and diagnostic status
Posttraumatic Stress Disorder Checklist for Civilians (PCL) | 1 month post baseline
  Parent PTSD severity and diagnostic status

SECONDARY OUTCOMES:
Center for Epidemiological Studies -Depression for Children (CES-DC) | 1 month post baseline
  Child depression severity and diagnostic status
Center for Epidemiological Studies -Depression (CES-D) | 1 month post baseline
  Parent depression severity and diagnostic status

CONTACTS AND LOCATIONS:
Overall Officials: Mark Burton, MA, Study Director — Case Western Reserve University
Locations (1):
- Akron children's Hospital, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No